CLINICAL TRIAL: NCT02193295
Title: Reversal of Lipid-Induced Insulin Resistance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 02029020997_a; R01DK135645 (NIH)
Record Dates: First submitted 2014-06-25; First posted 2014-07-17 (Estimated); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Insulin Resistance; NAFLD
Keywords: Weight Reduction; Caloric Restriction; Euglycemic Hyperinsulinemic Clamp; Magnetic Resonance Spectroscopy; PINTA
MeSH Terms: conditions — Insulin Resistance; Non-alcoholic Fatty Liver Disease; Weight Loss; Pinta | interventions — Caloric Restriction; Liver Extracts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Intervention (Experimental): Caloric Restriction to reverse lipid-induced insulin resistance.
  Interventions: Behavioral: Caloric Restriction
- Baseline Assessment of Hepatic Mitochondrial Fat Oxidation (Experimental): Tracer study to assess hepatic mitochondrial fat oxidation (PINTA).
  Interventions: Behavioral: Caloric Restriction

INTERVENTIONS:
Behavioral: Caloric Restriction — Dietary intervention to reduce lipid content in liver and muscle with minimal overall weight loss. Weekly visits for measurements of body weight, body composition, blood glucose and MRS measurements of liver and muscle lipid.
  Other Names: Dietary intervention to reduce lipid content in liver and muscle with minimal overall weight loss.

SUMMARY:
The purpose of this study is to examine whether weight reduction decreases intramyocellular (IMCL) and hepatic lipid content, and improves insulin sensitivity of muscle and fat tissue in people who are insulin resistant and have a family history of type 2 diabetes.

Hepatic mitochondrial oxidation will be assesses using a 3 hour triple tracer study (D7 glucose, 3-13C lactate and 13C4 beta-hydroxybutyrate).

DETAILED DESCRIPTION:
In this study, we will examine whether a small weight loss in lean, insulin-resistant offspring of type 2 diabetic patients will improve insulin resistance. The control group will consist of subjects matched for gender, age and body weight with no family history of diabetes. Before and after weight loss, rates of basal and insulin stimulated whole body glucose metabolism will be measured using [6,6-2H] glucose during a 3 hour basal period and a 4 hour euglycemic hyperinsulinemic (20 mU/m2-min) clamp. Rates of whole body lipolysis will be determined using [2H5] glycerol, localized rates of lipolysis will be measured using the microdialysis technique and muscle PI 3-kinase activity will be assessed in muscle biopsies. FFA metabolites (fatty acyl CoA, ceramides, diacylglycerol) will be measured in fat tissue collected from the abdominal subcutaneous fat cell depot. Body composition will be determined with bioelectrical impedance and whole body MRI; IMCL will be measured with MRS. Before and after weight loss, insulin secretion will be measured with the hyperglycemic clamp (as described under Day 2 Hyperglycemic Clamp).

Hepatic mitochondrial fat oxidation will be assessed in a separate study at baseline. Participants will be admitted to the Yale HRU at 7 AM after an overnight fast. An IV line will be placed in antecubital vein for tracer infusions and a retrograde IV line will be placed in a hand vein for blood collections. The hand will be warmed in a 'hot box' 37°C to approximate collection of 'arterial' blood samples. After collection of a baseline blood samples, infusions of 13C lactate (0.9 mM, 99% 13C, infusion rate: 8.7 micromol/(Kg-min)), D7glucose (25 mg/mL, 99% 13C, infusion rate: 0.84 mg/(m2-min)) and 13C-BHOB (2 mg/mL, 99%rate: 0.01 mg/(Kg-min)) will be started and continued for 180 minutes. During the final 20 minutes of this infusion period blood samples will be collected from the retrograde IV line. The infusion will then be discontinued the IV lines removed, and the participants will be served breakfast/lunch and discharged to home.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, sedentary, non-smoking and not taking any medications other than birth control pills.
* Hematocrit >35%
* Subjects will have no systemic or organ disease including diabetes.
* Subjects will have no history eating disorders.
* Women must be using a form of birth control (sexual abstinence, birth control pills, Norplant, IUD or condoms) and will be studied between day 0 and 7 of their menstrual cycle.
* Those who are taking birth control pills or have had a hysterectomy may be studied at any time.
* Physical activity will be assessed using a standard questionnaire with an activity index cut off at 2.3.

Exclusion Criteria:

* Any subject, who does not fit the inclusion criteria. Including history of eating disorders, any systemic and organ disease including diabetes.

Lactose intolerance Any blood count, clotting abnormalities HYpertriglyceridemeia (TG over 100 mg/dL)

* Hematocrit <35%.
* Women of childbearing potential, who are not using contraception (as mentioned above) or who are not abstinent.
* Subjects who have a regular exercise regimen will not be enrolled.
* Metal implants and/or body piercing, which cannot be removed before the MR studies.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2002-10 (Actual); Primary Completion 2034-10 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Improvements in insulin sensitivity | up to 6 months intervention to examine whether insulin sensitivity has improved significantly after the moderate weight reduction
  Insulin sensitivity will be assessed using the insulin/glucose clamp, liver and muscle fat will be measured using 1H magnetic resonance spectroscopy (MRS) and both results from the clamp and MRS compared to baseline values before the weight reduction intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kitt Petersen, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Magnetic Resonance Research Center (MRRC), New Haven, Connecticut
  - Yale Center for Clinical Investigation HRU, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No
Unidentified data will be provided to other investigators upon reasonable request after any publication of final data.